CLINICAL TRIAL: NCT03910439
Title: A Phase II Pilot Study of Avelumab in Combination With Hypofractionated Radiotherapy in Patients With Relapsed Refractory Multiple Myeloma
Brief Title: Avelumab in Combination With Hypofractionated Radiotherapy in Patients With Relapsed Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow/Insufficient accrual/COVID-19 pandemic
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190078; 19-C-0078
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Myeloma, Multiple; Myeloma-Multiple
Keywords: Monoclonal Antibody; Radiotherapy
MeSH Terms: conditions — Multiple Myeloma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Avelumab 800 mg intravenous (IV) every two weeks in combination with radiation therapy (Experimental): Avelumab 800 mg IV every two weeks in combination with radiation therapy
  Interventions: Biological: Avelumab; Radiation: External beam radiotherapy

INTERVENTIONS:
Biological: Avelumab — Avelumab 800 mg intravenous (IV) over 60 minutes (+/- 20 minutes) on days 1 and 15 of each 28-day cycle
  Other Names: MSB0010718C
Radiation: External beam radiotherapy — 5 gray (Gy) per fraction will be delivered on 5 consecutive treatment days for a total dose 25 Gy

SUMMARY:
Background:

Multiple myeloma is a cancer that forms from plasma cells which normally produce important immune response antibodies. It cannot be cured. Researchers hope the combination of radiation combined with the drug avelumab causes the immune system to kill myeloma cells more effectively.

Objective:

To see if avelumab given with radiation treatment helps treat multiple myeloma. Also to see if giving the treatments together is safe.

Eligibility:

People ages 18 and older with multiple myeloma that has come back after treatment and has spread to other parts of the body

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Possible tumor biopsy

Bone marrow testing: A needle will be stuck into the participants hipbone to take out a small amount of marrow.

Positron emission tomography (PET)/Computed tomography (CT) scan and magnetic resonance imaging (MRI): Participants will lie in a machine that takes pictures of the body.

Participants will get avelumab through an intravenous (IV). An IV is a small plastic tube put into an arm vein. They will get avelumab every 2 weeks for 2 doses. Then they will get radiation each day for 5 days. They will continue to get avelumab every 2 weeks as long as they do not have bad side effects and the treatment is helping their disease.

Participants will have blood and urine tests, bone marrow biopsies, scans, and X-rays repeated during the study.

Participants will have a follow-up visit 30 days after their last treatment dose. Then they will have visits every 3-6 months for up to 5 years....

DETAILED DESCRIPTION:
Background:

* Multiple Myeloma (MM) is a hematologic neoplasm of the plasma cells defined by an M- protein greater than or equal to 3.0 g/dL or bone marrow plasma cells greater than or equal to 10% and presence of end-organ disease.
* Although significant advances in treatment have been made in the past decade, MM remains incurable with median survivals of 5-8 years.
* While therapeutic strides have been made with approvals of immunomodulatory drugs (IMiDs), proteasome inhibitors, and monoclonal antibodies, treatment of relapsed refractory MM (RRMM) remains an unmet need for patients who have exhausted available therapies.
* Extramedullary plasmacytomas arising either from focal bone involvement or from hematogenous spread occur in 7-18% of newly diagnosed MM (NDMM) with an additional 6-20% in RRMM.
* Immune checkpoint inhibitors are being evaluated in combination regimens and evidence exists that radiation therapy (XRT) may synergize with immune checkpoint inhibitors.

Objectives:

- To assess the response rate of avelumab in combination with XRT (BavXRT) in RRMM patients with plasmacytomas or lytic lesions

Eligibility:

* Patients must have previously treated RRMM refractory to, ineligible for, or intolerant of available therapeutic regimens known to provide clinical benefit (e.g, immunomodulatory [IMiD], proteasome inhibitor, and anti-cluster of differentiation (CD)38 monoclonal antibody-based treatments).
* Presence of greater than or equal to 1 extramedullary plasmacytoma and/or lytic lesion amenable to XRT
* Age greater than or equal to 18 years
* Adequate organ function, and without serious comorbidity or disease (e.g., autoimmune disease), that would preclude concurrent systemic treatment or radiotherapy.

Design:

* Treatment will consist of a 4-week lead-in with avelumab, followed by concurrent XRT 5 gray (Gy) x 5 days). Monotherapy avelumab will continue indefinitely until progressive disease (PD) or unacceptable toxicity; 28-day cycles.
* Routine safety and MM-specific clinical labs will be assessed. Additional research bloods will be collected for evaluating immune-subsets, endosomes, and peripheral blood T cell repertoire prior to and following treatment (lead-in and prior to XRT, at disease re- evaluations at at time of response [i.e., complete remission (CR)/progressive disease (PD)]).
* Bone marrow biopsies will be evaluated for Programmed death-ligand 1 (PD-1)/ligand 1 (L1) expression, and B and T cell subsets using immunohistochemistry (IHC). Flow cytometry will also be used to evaluate stimulatory and inhibitory immune subsets along with endosomes. Standard clinical histopathology and flow cytometry will also be evaluated.
* Single arm, Simon minimax two-stage phase II trial design. The first stage will enroll 13 patients; if futility is not met, second stage will enroll another 14 patients to define the response rate to BavXRT in this population. Early stopping rules for safety will also be applied.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a documented diagnosis of multiple myeloma defined by the International Myeloma Working Group Criteria (IMWG)(3). Patients at initial diagnosis must have had a serum M-protein greater than or equal to 3 g/dL and/or bone marrow plasma cells greater than or equal to 10%, and at least one of the following:

  * Anemia: Hemoglobin less than or equal to10 g/dL, or
  * Renal failure: serum creatinine greater than or equal to 2.0 mg/dL, or
  * Hypercalcemia: Calcium (Ca) greater than or equal to10.5 mg/dL, or
  * Lytic bone lesions on X-ray, computed tomography (CT), or positron emission tomography (PET)/CT, or
  * greater than or equal to 2 focal lesions on spinal magnetic resonance imaging (MRI), or
  * greater than or equal to 60% bone marrow plasma cells, or
  * Involved/un-involved serum free light chain ratio greater than or equal to 100
* Have at least one extramedullary plasmacytoma or lytic lesion which at the discretion of the investigators is amenable to and clinically indicated for localized radiation therapy
* Must have Relapsed or Relapsed and Refractory Multiple Myeloma. Patients must have documented evidence of progressive disease (PD) as defined by the IMWG criteria on or after their last regimen and must have achieved a minimal response (MR) or better to at least one prior regimen. Definitions by the IMWG:

  * Relapsed and refractory: disease that is nonresponsive while on salvage therapy or progresses within 60 days of last therapy in patients who have achieved minor response (MR) or better
  * Relapsed: disease that progresses and requires the initiation of salvage therapy but does not meet criteria for either primary refractory or relapsed and refractory MM categories
* Patients must have been previously treated for MM and be refractory to, not a candidate for (ineligible), or intolerant of available therapeutic regimens known to provide clinical benefit including immunomodulatory (IMiD), proteasome inhibitor, and anti-cluster of differentiation (CD)38 monoclonal antibody-based treatments.
* Documented measurable disease within the 4 weeks prior to registration defined by any one of the following:

  * Monoclonal Bone marrow plasma cells greater than or equal to 5%
  * Serum monoclonal protein greater than or equal to 0.2 g/dl
  * Urine monoclonal protein >200 mg/24 hour
  * Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio
  * A measurable lesion on PET/CT or MRI
* Be greater than or equal to 18 years of age on day of signing informed consent

Note: The estimated 2017 US incidence of MM of patients under the age of 20 is 0.0%; therefore, children are excluded from enrollment in this study.

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate organ function as evidenced by the following laboratory parameters:

  * Absolute neutrophil count (ANC) greater than or equal to 1000 /mcL
  * Platelets greater than or equal to 75,000 / mcL
  * Hemoglobin greater than or equal to 8 g/dL (transfusions permitted)
  * Serum creatinine less than or equal to 1.5 X upper limit of normal (ULN) (except if due to myeloma)

OR

* Measured creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD- EPI) formula may be used to estimate CrCl/eGFR greater than or equal to 30 mL/min/1.73 m(2) for subject with creatinine levels > 1.5 X ULN
* Serum total bilirubin less than or equal to 1.5 X ULN OR Direct bilirubin less than or equal to ULN for patients with total bilirubin levels > 1.5 ULN (except if due to myeloma)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 X ULN (except if due to myeloma)

  * The effects of avelumab on the developing human fetus are unknown, however, given the known role of Programmed Cell Death Ligand 1 (PD-1)/Programmed death-ligand 1 (PD-L1) in maintaining the maternal/fetal tolerance, avelumab can be expected to have an adverse effect on pregnancy, including embryo-lethality. Women of child-bearing potential (WOCBP) and men must agree to use highly effective contraception (such as implants, injectables, combined oral contraceptives, intrauterine device (IUDs), sexual abstinence or vasectomised partner) prior to study entry and for the duration of study treatment, and for at least 30 days after the last dose of avelumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

* Negative serum or urine pregnancy test at screening for WOCBP.
* Ability of patient to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Patients with clinically unstable lesions (e.g., impending cord compression) where a delay in receiving radiation therapy (XRT) would be detrimental are not eligible
* Current or prior anti-cancer treatment prior to the first dose of avelumab as defined below:

  * Chemotherapy, targeted small molecule therapy, or other anti-cancer treatment not otherwise specified below within 2 weeks
  * Radiation therapy within 2 weeks
  * Anti-cancer monoclonal antibody (mAb) treatment within 4 weeks
  * Use of an investigational agent (e.g., biologic, drug, or other) within 4 weeks
  * Allogeneic stem cell transplant
* No autoimmune disease, as follows:

  * Active (acute or chronic) autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with type I diabetes, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment may be eligible.
  * History of serious autoimmune-related disorders including immune colitis, inflammatory bowel disease, pneumonitis, or pulmonary fibrosis whether drug- mediated or not.
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the patient in the judgment of the investigator:

  * Patients with a positive hepatitis B core antibody [HBcAb] and negative surface antigen (HBsAg) may be included if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable
  * Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
  * Known acquired immunodeficiency syndrome (AIDS). Controlled and stable human immunodeficiency virus (HIV) positivity is allowed
  * Prior organ transplantation including allogenic stem-cell transplantation
  * Clinically significant cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class III), or serious cardiac arrhythmia requiring medication. Mild arrhythmias, e.g. stable atrial fibrillation, may be allowed at the discretion of the investigator
  * Active infection requiring systemic therapy (minor infections may be allowed at the discretion of the investigator)
  * Known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the patient inappropriate for entry into the study.
* Persisting toxicity related to prior therapy (Grade > 1); however, alopecia, sensory neuropathy Grade less than or equal to 2, or other Grade less than or equal to 2 not constituting a safety risk based on investigator s judgment are acceptable.
* Vaccination with live vaccines within 4 weeks of the first dose of avelumab and while on study is prohibited (inactivated vaccines may be administered).
* Pregnant or lactating females. Because there is an unknown but potential risk for adverse events in nursing infants, on-study breastfeeding is not allowed.
* History of allergic reactions or hypersensitivity to avelumab or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (Grade greater than or equal to 3) unless felt to be in the best interests of the patient at the discretion of the investigator.
* Known additional malignancy that is symptomatic or requires active systemic treatment (at the discretion of the principal investigator (PI), exceptions may be made if in the best interest of the patient).
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0078.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.44 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as participants who experience a partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR) per International Myeloma Working Group Criteria (IMWG) 2016 criteria. Complete Response is defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. Stringent Complete Response is defined as complete response as noted previously plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow biopsy by immune-histochemistry. Partial Response is ≥50% reduction of serum M-protein plus reduction in 24 hour(h) urinary M-protein by ≥90% or to <200 mg per 24 h. Very Good Partial Response is serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 h.
Time Frame: up to end of study, an average of 11 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Proportion of participants
  Complete Response | 0 [0 to 0]
  Stringent Complete Response | 0 [0 to 0]
  Partial Response | 0 [0 to 0]
  Very Good Partial Response | 0 [0 to 0]

2. Secondary Outcome: Fraction of Participants Who Experience a Complete Response (CR) or Stringent Complete Response (sCR) Using the Study Treatment
Description: Response was assessed by the International Myeloma Working Group (IMWG) response criteria, 2016. Complete Response is defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. Stringent Complete Response is defined as complete response as noted previously plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow biopsy by immune-histochemistry.
Time Frame: up to end of study for individual patient, an average of 11 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Proportion of participants | 0 [0 to 0]

3. Secondary Outcome: Fraction of Participants Who Experience a Minimal Residual Disease Negative (MRDneg)Complete Response (CR) Using the Study Treatment
Description: Response was assessed by the International Myeloma Working Group Criteria (IMWG) 2016 criteria. Sustained MRDnegCR is defined as negativity in the marrow (next-generation flow (NGF) or next-generation sequencing (NGS), or both) and by imaging confirmed minimum of 1 year apart.
Time Frame: up to up to end of study for individual patient, an average of 11 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Proportion of participants | 0 [0 to 0]

4. Secondary Outcome: Percent Change in Aberrant Circulating Plasma Cells in the Peripheral Blood (PB) and Bone Marrow (BM) From Baseline
Description: Blood samples and bone marrow samples were taken from participants and processed by flow cytometry.
Time Frame: Baseline and up to end of study for individual patient, an average of 11 months
Measure: Mean (Full Range); unit: Percent change
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Percent change
  Peripheral blood at baseline | 0 [0 to 0]
  Bone marrow at baseline | 0 [0 to 0]
  Peripheral blood at end of study | 18 [-1 to 1000]
  Bone marrow at end of study | 55 [-0.01 to 1250]

5. Secondary Outcome: Percent Reduction in Size of On-irradiated Extramedullary Lesions
Description: Radiographic reduction in size of non-irradiated extramedullary lesions.
Time Frame: end of study
Population: This outcome measure was not evaluated due to study closure.
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Fluorodeoxyglucose (FDG) Avidity Positron-Emission Tomography/Computed Tomography (PET/CT) of Non-irradiated Extramedullary Lesions (Abscopal Effect) Compared to Baseline
Description: FDG avidity of extramedullary lesions.
Time Frame: End of study
Population: This outcome measure was not evaluated due to study closure.
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as those who progress or die without progression as failures, and censoring those who do not. Progressive disease was assessed by the 2016 International Myeloma Working Group (IMWG) response criteria and is an increase of 25% from lowest confirmed response value in one or more of the following criteria: Serum M-protein (absolute increase must be ≥0·5 g/dL); Serum M-protein increase ≥1 g/dL, if the lowest M component was ≥5 g/dL; Urine M-protein (absolute increase must be ≥200 mg/24 h); In patients without measurable serum and urine M-protein levels, the difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be >10 mg/dL).
Time Frame: End of study, an average of 11 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Months | 5.3 [2.5 to 7.1]

8. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Participants who are alive following enrollment and study treatment.
Time Frame: Enrollment through end of study, an average of 11 months
Measure: Number; unit: percentage of participants
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
percentage of participants | 100

9. Secondary Outcome: Number of Participants With Grade ≥1 Non-serious Adverse Events
Description: Grade ≥1 non-serious adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. Grade 1 is mild, Grade 2 is moderate, and Grade 3 is severe or medically significant.
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 4 days.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1: Grade 1 is mild.
- Grade 2: Grade 2 is moderate.
- Grade 3: Grade 3 is severe or medically significant.
Arm/Group | Grade 1 | Grade 2 | Grade 3
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Alanine aminotransferase increased | 1 | 1 | 0
  Alkaline aminotransferase increased | 1 | 0 | 0
  Arthralgia | 1 | 0 | 0
  Aspartate aminotransferase increased | 1 | 1 | 0
  Chest pain - cardiac | 0 | 1 | 0
  Eye disorders - Other, posterior vitreous detachment | 1 | 0 | 0
  Nausea | 1 | 0 | 0
  Pain | 1 | 1 | 0
  Rash maculo-papular | 1 | 0 | 0
  Skin infection | 1 | 0 | 0
  Syncope | 0 | 0 | 1
  Vomiting | 0 | 1 | 0

10. Secondary Outcome: Number of Participants Overall Best Response
Description: Response was assessed by the International Myeloma Working Group (IMWG) response criteria, 2016. Minimal Response is ≥25% but ≤49% reduction of serum M-protein and reduction in 24-h urine M-protein by 50-89%; in addition, if present at baseline, a ≥50% reduction in the size (SPD) of soft tissue plasmacytomas is also required. Stable Disease is not meeting criteria for complete response, very good partial response, partial response, minimal response, or progressive disease. And Progressive Disease is appearance of a new lesion(s), ≥50% increase from nadir in sum of the products of diameters (SPD) of >1 lesion, or ≥50% increase in the longest diameter of a previous lesion >1 cm in short axis; ≥50% increase in circulating plasma cells (minimum of 200 cells per microliter (μL) if this is the only measure of disease.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Participants
  Minimal Response | 1
  Stable Disease | 2
  Progressive Disease | 1

11. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 4 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 4 days.
Arm/Group | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Avelumab 800 mg Intravenous (IV) Every Two Weeks in Combination With Radiation Therapy (N=4)
Alanine aminotransferase increased (Investigations) | 1 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Chest pain - cardiac (Musculoskeletal and connective tissue disorders) | 1 (1)
Eye disorders - Other, posterior vitreous detachment (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03910439/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03910439/ICF_001.pdf